CLINICAL TRIAL: NCT00606801
Title: Galantamine Effects on Cognitive Function in Abstinent Cocaine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0706002768; P50DA009241 (NIH); B Rounsaville (Other: Principal Investigator of P50 grant)
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Cocaine Abuse
Keywords: cognitive enhancers; Nootropic Agents
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Galantamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine 8 mg/day (Active Comparator): Galantamine 8 mg/day
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Galantamine — Galantamine 8 mg/day
  Other Names: Nivalin,; Razadyne,; Razadyne ER,; Reminyl,; Lycoremine
  Arms: Galantamine 8 mg/day
Drug: placebo — sugar pill
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
To evaluate galantamine's effects on cognitive performance in abstinent cocaine users. Galantamine, a medication approved for treatment of Alzheimer's disease, is an acetylcholine esterase inhibitor. Galantamine also directly potentiates nicotine receptors. Both of these effects may result in improved cognitive performance in a group of subjects known to have impaired performance in various cognitive tasks.

DETAILED DESCRIPTION:
Galantamine, compared to placebo, will improve cognitive performance in abstinent cocaine users. The cognitive performance will be measured with the Stroop test and 3 Cambridge Neuropsychological Test Automated Battery (CANTAB) tests: Paired Associate Learning (PAL), Delayed Pattern Recognition Memory (PRM),and Rapid Visual Information Processing (RVIP). Performance on these tests has been shown to be impaired in abstinent cocaine users, compared to healthy controls.

Galantamine, compared to placebo, will not be associated with any significant changes in mood. Monitoring of mood will be achieved with 3 mood scales: 1) Center for Epidemiologic Studies Depression (CES-D) scale, Positive and Negative Affect Schedule (PANAS) and the Profile of Mood States (POMS).

Currently this study is completed, Patients are no longer being enrolled. There were 28 completers. This study has been published.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, between the ages 21 and 50
* Fulfill criteria for past cocaine dependence
* No cocaine use for the past 30 days
* No other current dependence or abuse of other drugs or alcohol
* No current medical problems and normal ECG
* Not pregnant,nor breast feeding,
* Using acceptable birth control methods.

Exclusion Criteria:

* Current major psychiatric illness including mood, psychotic or anxiety disorders
* History of major medical illnesses; including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal impairment and cardiac rhythm disturbances
* Use of other medications including,drugs that slow heart rate
* Known allergy to galantamine

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University Associate Professor
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Abstinent cocaine users recruited from 2007 to 2009 using word of mouth, fliers, and newspaper advertisements. This was an outpatient study conducted in a Yale University & Veteran Affairs substance abuse research clinic.
Pre-assignment Details: 55 subjects were screened. 21 subjects were excluded. (Not meeting inclusion criteria n=19, declined to participate n=2). These 34 subjects were then assigned to treatment groups. Prior to the 1st day of intervention, subjects underwent an adaptation session where they were familiarized with study procedures, and baseline measures were obtained.
Groups:
- Placebo: Placebo given for 10 days.
- Galantamine 8 mg/Day: Galantamine 8 mg/day given for 10 days.
Period: Adaptation
Arm/Group | Placebo | Galantamine 8 mg/Day
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Intervention
Arm/Group | Placebo | Galantamine 8 mg/Day
Started | 17 | 17
Completed | 14 | 14
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine 8 mg/Day | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (5.9) | 42.7 (6.3) | 42.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - RVIP Reaction Time
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the RVIP, subjects must detect either odd or even 3 digit sequences appearing in a box in a pseudo-random order at 100 digits per minute. Reaction time (RT) to correct answers was measured.
Time Frame: Baseline, Day 5 and Day 10
Population: There were a total of 28 completers, 14 for each treatment group. However, CANTAB data was not stored on the hard drive for one subject in the Galantamine group.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Placebo: Measures on placebo group.
- Galantamine: Measures on Galantamine group.
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
milliseconds
  Baseline | 407.7 (92.3) | 476.8 (119.3)
  Day 5 | 427.4 (35.3) | 379.2 (71.7)
  Day 10 | 433.3 (123.6) | 386.9 (82.9)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; A mixed-effect, repeated-measures model using main effect terms of treatment (placebo or galantine) and time (day of measurement). Interaction of main effects were also analyzed, with a random effect for participant. Given the hypothesis generating nature of the study, values of p<0.05 were considered statistically significant based on two-tailed tests. Significant interactions were followed by Bonferroni post hoc pairwise comparisons; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis

2. Primary Outcome: Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - RVIP Total Hits
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the RVIP, subjects must detect either odd or even 3 digit sequences appearing in a box in a pseudo-random order at 100 digits per minute. The total hits were measured
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hits
Groups:
- Placebo: Measures on the placebo group.
- Galantamine: Measures on the Galantamine group.
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
hits
  Baseline | 16.7 (3.6) | 14.8 (4.7)
  Day 5 | 18.0 (5.0) | 16.9 (5.4)
  Day 10 | 18.0 (6.8) | 19.7 (4.3)
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis

3. Primary Outcome: Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - RVIP Total Correct Rejections
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the RVIP, subjects must detect either odd or even 3 digit sequences appearing in a box in a pseudo-random order at 100 digits per minute. The number of correct rejections was measured.
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct rejections
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
correct rejections
  Baseline | 247.2 (13.7) | 242.4 (15.5)
  Day 5 | 217.6 (16.9) | 247.9 (12.9)
  Day 10 | 248.2 (23.7) | 253.9 (12.6)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

4. Primary Outcome: Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - RVIP A' (Sensitivity to Target Sequences)
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the RVIP, subjects must detect either odd or even 3 digit sequences appearing in a box in a pseudo-random order at 100 digits per minute. A' is a measure of sensitivity to target sequences and it reflects probabilities of hits and false alarms to provide a score of sensitivity to the target regardless of response tendency. The scores range from 0 (bad) to 1 (good).
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sensitivity index
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
sensitivity index
  Baseline | 0.89 (0.04) | 0.87 (0.07)
  Day 5 | 0.90 (0.07) | 0.90 (0.07)
  Day 10 | 0.90 (0.10) | 0.92 (0.04)
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

5. Primary Outcome: Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - RVIP B' (Strength to Detect to Target Sequences)
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the RVIP, subjects must detect either odd or even 3 digit sequences appearing in a box in a pseudo-random order at 100 digits per minute. B reflects the probability of hits and false alarms to provide a measure of the participants tendency to respond regardless of whether the target sequence is presented. The scores range from -1 to +1 with scores near +1 indicative of a subject that gave few false alarms.
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: specificity index
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
specificity index
  Baseline | .88 (.18) | .88 (.25)
  Day 5 | .82 (.22) | .91 (.11)
  Day 10 | .85 (.25) | .88 (.14)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5, Mixed Models Analysis

6. Primary Outcome: Paired Associate Learning (PAL) - Stages Complete
Description: Rapid Visual Processing test (RVIP) is a measure of sustained attention with a small working memory component that is sensitive to cholinergic enhancers. In the Paired Associate Learning (PAL) task, boxes are displayed on the screen and are opened in a random order. One or more of the boxes will contain a pattern. After the subjects have seen the patterns behind each box, the patterns are then displayed in the middle of the screen, one at a time, and the subject must touch the box where the pattern was originally located. An error will cause the test to open the boxes again to remind the subject of their locations. The number of boxes with patterns increases throughout the test. The stages completed and number of errors are measures of interest.
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: completed stages
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
completed stages
  Baseline | 4.8 (.4) | 4.9 (.4)
  Day 5 | 4.9 (.4) | 4.9 (.4)
  Day 10 | 4.9 (.4) | 4.9 (.4)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis

7. Primary Outcome: Paired Associate Learning (PAL) - Mean Errors
Description: as for outcome 6
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
errors
  Baseline | 31.1 (22.3) | 25.6 (16.5)
  Day 5 | 23.6 (17.7) | 18.1 (11.5)
  Day 10 | 17.7 (16.6) | 16.8 (13.7)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis

8. Primary Outcome: Pattern Recognition Memory (PRM) - Response Time for Correct Answers
Description: In the PRM, the subject is presented with a series of 12 visual patterns, one at a time, in the center of the screen. These patterns are designed so that they cannot easily be given verbal labels. In the recognition phase, the subject is required to choose between a pattern they have already seen and a novel pattern. The time to correct answer was measured.
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
milliseconds
  Baseline | 2357 (526) | 2439 (685)
  Day 5 | 2092 (573) | 2092 (522)
  Day 10 | 1995 (479) | 1889 (364)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis

9. Primary Outcome: Pattern Recognition Memory (PRM) - Number Correct Answers
Description: Pattern Recognition Memory (PRM) tests visual pattern recognition memory in a two choice forced discrimination paradigm. 12 visual patterns are presented, then the subject must choose between each of these patterns and a novel pattern. The number of correct responses are measured.
Time Frame: Baseline, Day 5 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number correct answers
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 14 | 13
number correct answers
  Baseline | 20.8 (3.2) | 20.2 (2.5)
  Day 5 | 14.9 (2.9) | 20.6 (2.5)
  Day 10 | 21.0 (2.9) | 20.7 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis

10. Secondary Outcome: Performance on the Sustained Attention to Response Task (SART) - Number of Errors on NoGo Trials
Description: The SART is a Go / NoGo task measuring the ability to activate or inhibit responses. In this 4.5 minute task, 225 single digits (25 × 9 digits) were presented on a computer monitor. Each digit was presented for 250 ms, and was immediately followed by a mask for 900 ms. The mask consists of a ring with a diagonal cross in the center. Subjects were instructed to press a spacebar to every digit except the 3, and to give equal importance to speed and accuracy. Responses were allowed during the presentation of both the digit and mask. The digits were presented in a different random order for each subject. There were 18 practice trials, containing 2 no-response targets (3s). For the Go/NoGo task, response inhibition was measured as the number of errors on the no- Go trials, with low errors indicating better response inhibition.
  Complete data for 3 subjects in the Placebo group, and for 1 subject in the galantamine group were not capture do to experimenter and computer errors.
Time Frame: Baseline, Day 5 and Day 10
Population: Participants analyzed are those that completed the treatment phase.
Measure: Mean (Standard Deviation); unit: number of errors
Groups:
- Placebo: Measures in placebo group.
- Galantamine: Measures in galantamine group.
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 11 | 13
number of errors
  Baseline | 12.8 (6.4) | 13.1 (5.8)
  Day 5 | 10.7 (6.5) | 10.2 (7.9)
  Day 10 | 11.8 (7.7) | 12.2 (8.2)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9, Mixed Models Analysis

11. Secondary Outcome: Performance on the Sustained Attention to Response Task (SART)- Number of Errors on Go Trials
Description: The SART is a Go / NoGo task measuring the ability to activate or inhibit responses. In this 4.5 minute task, 225 single digits (25 × 9 digits) were presented on a computer monitor. Each digit was presented for 250 ms, and was immediately followed by a mask for 900 ms. The mask consists of a ring with a diagonal cross in the center. Subjects were instructed to press a spacebar to every digit except the 3, and to give equal importance to speed and accuracy. Responses were allowed during the presentation of both the digit and mask. The digits were presented in a different random order for each subject. There were 18 practice trials, containing 2 no-response targets (3s). The number of errors on Go trials reflected the response activation function, with fewer errors indicating greater response activation.
  Complete data for 3 subjects in the Placebo group, and for 1 subject in the galantamine group were not capture do to experimenter and computer errors.
Time Frame: Baseline, Day 5 and Day 10
Population: Participants analyzed are those that completed the treatment phase.
Measure: Mean (Standard Deviation); unit: the number of errors
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 11 | 13
the number of errors
  Baseline | 14.6 (16.8) | 7.2 (7.4)
  Day 5 | 12.0 (19.1) | 3.8 (4.1)
  Day 10 | 10.6 (10.6) | 5.1 (7.4)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8, Mixed Models Analysis

12. Secondary Outcome: Performance on the Sustained Attention to Response Task (SART)- Mean Reaction Time for Correct Press on Go Trial
Description: The SART is a Go / NoGo task measuring the ability to activate or inhibit responses. In this 4.5 minute task, 225 single digits (25 × 9 digits) were presented on a computer monitor. Each digit was presented for 250 ms, and was immediately followed by a mask for 900 ms. The mask consists of a ring with a diagonal cross in the center. Subjects were instructed to press a spacebar to every digit except the 3, and to give equal importance to speed and accuracy. Responses were allowed during the presentation of both the digit and mask. The digits were presented in a different random order for each subject. There were 18 practice trials, containing 2 no-response targets (3s).
  For the Go trial, the reaction time reflected the response activation function, faster reaction time indicating greater response activation.
  Complete data for 3 subjects in the Placebo group, and for 1 subject in the galantamine group were not capture do to experimenter and computer errors.
Time Frame: Baseline, Day 5 and Day 10
Population: Participants analyzed are those that completed the treatment phase.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 11 | 13
milliseconds
  Baseline | 399.7 (79.7) | 375.3 (88.5)
  Day 5 | 405.4 (81.7) | 382.6 (79.9)
  Day 10 | 411.1 (74.2) | 357.8 (109.7)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5, Mixed Models Analysis

13. Secondary Outcome: Performance on the Modified Stroop Task (Cocaine-Stroop)- Reaction Time
Description: The Cocaine-Stroop task measures attention capture (attentional bias) secondary to cocaine cues; (Stroop effect - calculated as the difference between mean RT on cocaine words and mean RT on control words). Subjects completed 2 counterbalanced blocks (150 trials per block). One block contained 15 cocaine words and neutral words in a mixed order. The other block contained 15 control words matched in length and frequency to cocaine words, and a different set of neutral words. Subjects were required to indicate the colors in which the words were written as quickly and accurately as possible. Reaction times for identification of word color was measured. In addition, the difference in RT to words following cocaine and control words were measured (carry-over effect). Complete data for 3 participants (2 placebo and 1 galantamine) were not capture due to experimenter and computer errors.
Time Frame: Baseline, Day 5 and Day 10
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 12 | 13
milliseconds
  Baseline | 722 (117) | 771 (136)
  Day 5 | 734 (126) | 742 (145)
  Day 10 | 748 (159) | 698 (106)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

14. Secondary Outcome: Performance on the Modified Stroop Task (Cocaine-Stroop)- Stroop Effect
Description: as for outcome 13
Time Frame: Baseline, Day 5 and Day 10
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 12 | 13
milliseconds
  Baseline | 10.5 (66.2) | -13.1 (137.6)
  Day 5 | -19.7 (87.6) | 19.6 (149.3)
  Day 10 | -61.5 (183.9) | -33.7 (133.2)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis

15. Secondary Outcome: Performance on the Modified Stroop Task (Cocaine-Stroop)- Carry-over Effect
Description: as for outcome 13
Time Frame: Baseline, Day 5 and Day 10
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Galantamine
Number analyzed (Participants) | 12 | 13
milliseconds
  Baseline | 32.4 (95.5) | 13.4 (131.9)
  Day 5 | 43.5 (131.2) | 32.1 (96.2)
  Day 10 | -29.8 (179.6) | 18.6 (110.5)
Statistical Analysis 1: Comparison: Placebo vs Galantamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.50, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Galantamine 8 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Relatively low medication dose and short duration of treatment. Multiple cognitive tests and outcome measures increase probability of Type 1 errors. Absence of non-addicted controls limits determination of a unique effect in abstinent users.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No